CLINICAL TRIAL: NCT00919113
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group Evaluation of the Effectiveness and Safety of Uracyst® Compared to Inactive Control in Subjects With Interstitial Cystitis/Painful Bladder Syndrome
Brief Title: Efficacy and Safety Study of Uracyst to Treat Interstitial Cystitis/Painful Bladder Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UR08004
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
Keywords: Bladder Pain; GAG replacement therapy; IC/PBS
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Chondroitin Sulfates; Buffers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8 weekly bladder instillations of Uracyst (Experimental): 20 mL Uracyst (2% sodium chondroitin sulfate) per instillation; 8 instillations over a 7-week period
  Interventions: Drug: 2% sodium chondroitin sulfate
- 8 weekly bladder instillations of inactive control (Placebo Comparator): 20 mL inactive control buffer (phosphate-buffered saline); 8 instillations over a 7-week period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2% sodium chondroitin sulfate — Weekly 20 mL Intravesical instillation
  Other Names: Uracyst
  Arms: 8 weekly bladder instillations of Uracyst
Drug: Placebo — The identical buffer used in Uracyst for the same administration
  Other Names: buffer
  Arms: 8 weekly bladder instillations of inactive control

SUMMARY:
A new device for interstitial cystitis is compared to inactive control to determine if it is safe and effective. The study lasts approximately 7 weeks with a 19-week follow-up period.

DETAILED DESCRIPTION:
Multi-center, randomized, double-blind, parallel, 8 weekly instillations over a 7-week period with post-treatment follow-up for an additional 19 weeks for a total study length of 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are a female, 18 years or older
* Have been diagnosed with IC/PBS
* Are willing to provide written informed consent and authorization to disclose after being fully informed of the risks of participation

Exclusion Criteria:

* Are lactating females
* Have previously received investigational products or devices within 30 days of screening
* Have previously received Uracyst
* Are currently receiving therapy with Interstim®
* Have any other condition/disease which, in the opinion of the investigator, could compromise subject safety or confound the interpretation of study results
* Are unable or unwilling to comply with protocol requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Hill, PharmD, MBA, Study Director — Watson Laboratories, Inc.
Locations (20):
- United States (20):
  - Boulder, Colorado
  - Denver, Colorado
  - Farmington, Connecticut
  - Plantation, Florida
  - Wellington, Florida
  - Columbus, Georgia
  - Coeur d'Alene, Idaho
  - Evanston, Illinois
  - Melrose Park, Illinois
  - Royal Oak, Michigan
  - Las Vegas, Nevada
  - Englewood, New Jersey
  - Sewell, New Jersey
  - Woodlane, New Jersey
  - Albany, New York
  - Poughkeepsie, New York
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Mountlake Terrace, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Uracyst: 2% sodium chondroitin sulfate
- Placebo: identical buffer
Period: Overall Study
Arm/Group | Uracyst | Placebo
Started | 50 | 48
Received Uracyst | 49 (One subject was misrandomized. Actual treatment was used for Demographic and Safety analysis.) | 0
Received Placebo | 0 | 49 (One subject was misrandomized. Actual treatment was used for Demographic and Safety analysis.)
Completed | 41 | 40
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uracyst | Placebo | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 4 | 4 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 44.4 (14.6) | 46.8 (14.1) | 45.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98

OUTCOME MEASURES:

1. Primary Outcome: Global Response Assessment (GRA) Responders at Week 11.
Description: subjects that indicated "markedly improved" or "moderately improved" on the GRA, LOCF
Time Frame: at week 11
Population: Efficacy analysis performed according to randomized treatment.
Measure: Number; unit: participants
Arm/Group | Uracyst | Placebo
Number analyzed (Participants) | 50 | 48
participants | 19 | 15

2. Secondary Outcome: Interstitial Cystitis Symptom Index (ICSI) Responders at Week 11.
Description: Subjects that exhibited at least a 30% improvement from baseline in their total ICSI score, LOCF
Time Frame: at week 11
Population: Efficacy analysis performed according to randomized treatment.
Measure: Number; unit: participants
Arm/Group | Uracyst | Placebo
Number analyzed (Participants) | 50 | 48
participants | 23 | 18

ADVERSE EVENTS:
Groups:
- Uracyst: 2% sodium chondroitin sulfate
  One subject was misrandomized. Actual treatment was used for Demographic and Safety analysis.
- Placebo: identical buffer
  One subject was misrandomized. Actual treatment was used for Demographic and Safety analysis.
Arm/Group | Uracyst | Placebo
Serious Adverse Events (participants affected / at risk) | 1/49 | 2/49
Other Adverse Events (participants affected / at risk) | 21/49 | 18/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uracyst (N=49) | Placebo (N=49)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Uracyst (N=49) | Placebo (N=49)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Dysuria (Renal and urinary disorders) | 6 | 4
Headache (Psychiatric disorders) | 1 | 6
Nausea (Gastrointestinal disorders) | 4 | 3
Cystitis Interstitial (Renal and urinary disorders) | 2 | 4
Urinary Tract Infection (Renal and urinary disorders) | 4 | 2
Bladder Pain (Renal and urinary disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less